CLINICAL TRIAL: NCT04331873
Title: Confirming Proper Replacement of Dislodged Gastrostomy Tubes in Pediatric Patients: Can we Replace Contrast Injection With Ultrasound
Brief Title: Confirming Proper Replacement of Dislodged Gastrostomy Tubes in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Le Bonheur Children's Hospital (Other)
Responsible Party: Principal Investigator, Cailin Frank, DO, Pediatric Emergency Medicine Fellow, University of Tennessee
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-06455-XP
Record Dates: First submitted 2019-04-15; First posted 2020-04-02 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Gastrostomy Tube Site Complication; Gastrostomy Complications
Keywords: gastrostomy; dislodged
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound (Experimental): An ultrasound will be obtained to evaluate placement of the gastrostomy tube prior to obtaining the standard contrast injection
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — An ultrasound will be obtained prior to obtaining the standard contrast injection to determine if this imaging modality is equivocal.
  Other Names: US

SUMMARY:
The purpose of this study is to evaluate if ultrasound can be used effectively to confirm location of gastrostomy tube (G-tube) placement in place of a study in which contrast is flushed through the G-tube and placement is checked with X-ray. A G-tube is a tube inserted through the abdomen and delivers nutrition directly into the stomach.

DETAILED DESCRIPTION:
The purpose of this study is to determine if ultrasound is a safe and reliable way to confirm the proper placement of a dislodged gastrostomy tube in a pediatric emergency department.

In the case of emergent replacement of dislodged gastrostomy tubes, the emergency department currently obtains a contrast injection of the gastrostomy tube to confirm proper replacement in patients who recently had gastrostomy surgically placed or those who require dilation/have difficult replacement as per the pediatric surgery protocol. In this study, an ultrasound (US) will be obtained by an US technician to assess if the gastrostomy tube is in the proper location. Once this study has been obtained, the patient will undergo the typical contrast injection of the gastrostomy tube to confirm placement. The sensitivity and specificity of ultrasound to the current gold standard of contrast injection will be compared.

Ultrasound (US) has the benefit of having no radiation exposure for the patient. In patients anticipated to have multiple emergency department visits a year for gastrostomy complications, using ultrasound as opposed to contrast injection may make a significant impact on accumulated radiation exposure.

The patient population will be composed of children ages 0 to 21 years that visit Le Bonheur Children's Hospital Emergency Department (Memphis, TN) for replacement of a dislodge gastrostomy tube who require contrast injection to confirm proper replacement. Once it is determined that imaging is needed to confirm replacement, the patient and legally authorized representative (LAR) will be consented for the study. The determination for contrast injection is made per protocol when gastrostomy was placed within the last 3 months or when a difficult replacement occurs (i.e. one requiring stoma dilation). A procedure checklist will be used for the provider to complete for the procedure that can be used to better evaluate the amount of attempts made to replace the tube and different methods used prior to decision to pursue contrast injection.

The LAR's will be consented for the study once they are in their private exam room in the ER. Consent, and assent when applicable, will be obtained for the study as well as discussion of risks of improper gastrostomy placement and it's risk of infection. However, this will not be deviating from the current standard of care for emergent gastrostomy replacement.

When patient goes to the radiology department, they will have an US performed by US technician who will inject Pedialyte solution through the gastrostomy and visualize fluid entering the stomach in sagittal and transverse views. These ultrasound images will not have any effect on the patient's ER course in real time and will be read by the attending radiologist the following day. Furthermore, the risk of Pedialyte injection into an improperly placed gastrostomy tube has already been discussed with pediatric surgery and radiology and is determined to be of no risk of harm to the patient as any misplaced tube would require confirmation with contrast injection at this point in time. The patient will then have contrast injection performed as per the standard of care to confirm placement and then will return to their ER exam room for further management during their visit based on the results of their contrast injection study.

ELIGIBILITY:
Inclusion Criteria:

* Dislodged gastrostomy tube requiring contrast injection to confirm proper gastrostomy replacement

Exclusion Criteria:

* No ultrasound technician present in hospital
* Non-functioning ultrasound equipment (e.g. due to hardware issues)

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Confirmation of gastrostomy tube placement | This procedure is brief (<5-10 minutes) and will be performed after gastrostomy tube replacement prior to the patient having the gold standard contrast injection performed before returning to their exam room. This should take no more than one hour
  Ultrasound will be obtained in addition to contrast injection to determine gastrostomy tube placement

CONTACTS AND LOCATIONS:
Overall Officials: Rudy A Kink, MD, Study Director — Le Bonheur Children's Hospital
Locations (1):
- LeBonheur Children's Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dookhoo L, Mahant S, Parra DA, John PR, Amaral JG, Connolly BL. Peritonitis following percutaneous gastrostomy tube insertions in children. Pediatr Radiol. 2016 Sep;46(10):1444-50. doi: 10.1007/s00247-016-3628-5. Epub 2016 May 12. PMID 27173980
- [Background] Myatt TC, Medak AJ, Lam SHF. Use of Point-of-Care Ultrasound to Guide Pediatric Gastrostomy Tube Replacement in the Emergency Department. Pediatr Emerg Care. 2018 Feb;34(2):145-148. doi: 10.1097/PEC.0000000000001400. PMID 29346232
- [Background] Saavedra H, Losek JD, Shanley L, Titus MO. Gastrostomy tube-related complaints in the pediatric emergency department: identifying opportunities for improvement. Pediatr Emerg Care. 2009 Nov;25(11):728-32. doi: 10.1097/PEC.0b013e3181bec847. PMID 19864965
- [Background] Showalter CD, Kerrey B, Spellman-Kennebeck S, Timm N. Gastrostomy tube replacement in a pediatric ED: frequency of complications and impact of confirmatory imaging. Am J Emerg Med. 2012 Oct;30(8):1501-6. doi: 10.1016/j.ajem.2011.12.014. Epub 2012 Feb 4. PMID 22306396
- [Background] Tsujimoto H, Tsujimoto Y, Nakata Y, Akazawa M, Kataoka Y. Ultrasonography for confirmation of gastric tube placement. Cochrane Database Syst Rev. 2017 Apr 17;4(4):CD012083. doi: 10.1002/14651858.CD012083.pub2. PMID 28414415
- [Background] Wu TS, Leech SJ, Rosenberg M, Huggins C, Papa L. Ultrasound can accurately guide gastrostomy tube replacement and confirm proper tube placement at the bedside. J Emerg Med. 2009 Apr;36(3):280-4. doi: 10.1016/j.jemermed.2007.11.064. Epub 2008 Jul 9. PMID 18614327
- [Background] Zamora IJ, Fallon SC, Orth RC, Kim ME, Brandt ML, Lopez ME, Wesson DE, Rodriguez JR. Overuse of fluoroscopic gastrostomy studies in a children's hospital. J Surg Res. 2014 Aug;190(2):598-603. doi: 10.1016/j.jss.2014.05.010. Epub 2014 May 9. PMID 24909868
- [Result] Berman L, Hronek C, Raval MV, Browne ML, Snyder CL, Heiss KF, Rangel SJ, Goldin AB, Rothstein DH. Pediatric Gastrostomy Tube Placement: Lessons Learned from High-performing Institutions through Structured Interviews. Pediatr Qual Saf. 2017 Feb 23;2(2):e016. doi: 10.1097/pq9.0000000000000016. eCollection 2017 Mar-Apr. PMID 30229155
- [Result] Bhambani S, Phan TH, Brown L, Thorp AW. Replacement of Dislodged Gastrostomy Tubes After Stoma Dilation in the Pediatric Emergency Department. West J Emerg Med. 2017 Jun;18(4):770-774. doi: 10.5811/westjem.2017.3.31796. Epub 2017 Apr 19. PMID 28611900
- [Result] Church JT, Speck KE, Jarboe MD. Ultrasound-guided gastrostomy tube placement: A case series. J Pediatr Surg. 2017 Jul;52(7):1210-1214. doi: 10.1016/j.jpedsurg.2017.03.061. Epub 2017 Apr 2. PMID 28408076
- [Result] Chenaitia H, Brun PM, Querellou E, Leyral J, Bessereau J, Aime C, Bouaziz R, Georges A, Louis F; WINFOCUS (World Interactive Network Focused On Critical Ultrasound) Group France. Ultrasound to confirm gastric tube placement in prehospital management. Resuscitation. 2012 Apr;83(4):447-51. doi: 10.1016/j.resuscitation.2011.11.035. Epub 2011 Dec 29. PMID 22209831
- [Result] Correa JA, Fallon SC, Murphy KM, Victorian VA, Bisset GS, Vasudevan SA, Lopez ME, Brandt ML, Cass DL, Rodriguez JR, Wesson DE, Lee TC. Resource utilization after gastrostomy tube placement: defining areas of improvement for future quality improvement projects. J Pediatr Surg. 2014 Nov;49(11):1598-601. doi: 10.1016/j.jpedsurg.2014.06.015. Epub 2014 Aug 8. PMID 25475801